CLINICAL TRIAL: NCT04825821
Title: A Prospective Pilot Study Comparing Incidence and Characteristics of Cesarean Scar Defects After Uterine Closure by Double-layer Barbed or Smooth Suture
Brief Title: Cesarean Scar Defects After Uterine Closure by Double-layer Barbed or Smooth Suture
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: BARB-CSCAR
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Isthmocele; Uterine Scar Defects; Cesarean Section Complications; Uterine Niche
Keywords: Uterine scar defects; Uterine niche; Isthmocele

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low transverse hysterotomy closed by double-layer unidirectional barbed suture: Patients who had undergone cesarean section during which the low transverse hysterotomy was closed by double-layer unidirectional barbed suture
  Interventions: Procedure: Clinical and ultrasonographic assessment
- Low transverse hysterotomy closed by conventional double-layer smooth suture: Patients who had undergone cesarean section during which the low transverse hysterotomy was closed by conventional double-layer smooth suture
  Interventions: Procedure: Clinical and ultrasonographic assessment

INTERVENTIONS:
Procedure: Clinical and ultrasonographic assessment — Routinely assessment by objective examination and transvaginal ultrasonographic scan 6, 12, and 24 months after the surgical procedures

SUMMARY:
Late sequelae of a cesarean section related to a uterine scar defects include gynecological symptoms and obstetric complications. The aim of this study was to evaluate the incidence and characteristics of cesarean scar defects after uterine closure by double-layer barbed suture.

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent elective cesarean section at ≥ 37 weeks of gestation

Exclusion Criteria:

* Patients who underwent concomitant surgical procedures during the cesarean section (i.e., tubal sterilization);
* Patients who underwent a previous abdominal surgery (with exception of appendectomy) including a cesarean section or other laparotomic/laparoscopic uterine surgical procedure (i.e., myomectomy);
* Patients who had a previous diagnosis of Mullerian uterine anomalies elective cesarean for the second time or after uterine surgery;
* Patients who had evidence of PAS disorders or placenta previa.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent elective cesarean section at ≥37 weeks of gestation
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of uterine scar defects | 6 months after the cesarean section
  Number of simple and complex uterine scar defects is evaluated by transvaginal ultrasound
Number of uterine scar defects | 12 months after the cesarean section
  Number of simple and complex uterine scar defects is evaluated by transvaginal ultrasound
Number of uterine scar defects | 24 months after the cesarean section
  Number of simple and complex uterine scar defects is evaluated by transvaginal ultrasound

SECONDARY OUTCOMES:
Residual myometrium thickness (RMT), depth, width and length of uterine scar defects | 6 months after the cesarean section
  RMT, depth, width, and length are evaluated by transvaginal ultrasound
Residual myometrium thickness (RMT), depth, width and length of uterine scar defects | 12 months after the cesarean section
  RMT, depth, width, and length are evaluated by transvaginal ultrasound
Residual myometrium thickness (RMT), depth, width and length of uterine scar defects | 24 months after the cesarean section
  RMT, depth, width, and length are evaluated by transvaginal ultrasound
Number of patients with postmenstrual spotting | 6 months after the cesarean section
  Number of patients with postmenstrual spotting is evaluated by medical interview
Number of patients with postmenstrual spotting | 12 months after the cesarean section
  Number of patients with postmenstrual spotting is evaluated by medical interview
Number of patients with postmenstrual spotting | 24 months after the cesarean section
  Number of patients with postmenstrual spotting is evaluated by medical interview
Number of patients with dysmenorrhea | 6 months after the cesarean section
  Number of patients with dysmenorrhea is evaluated by medical interview with VAS (visual analogue scale)
Number of patients with dysmenorrhea | 12 months after the cesarean section
  Number of patients with dysmenorrhea is evaluated by medical interview with VAS (visual analogue scale)
Number of patients with dysmenorrhea | 24 months after the cesarean section
  Number of patients with dysmenorrhea is evaluated by medical interview with VAS (visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Barra, MD, Principal Investigator — IRCCS Ospedale Policlinico San Martino
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agarwal S, D'Souza R, Ryu M, Maxwell C. Barbed vs conventional suture at cesarean delivery: A systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2021 Jun;100(6):1010-1018. doi: 10.1111/aogs.14080. Epub 2021 Feb 5. PMID 33404082
- [Background] Alessandri F, Evangelisti G, Centurioni MG, Gustavino C, Ferrero S, Barra F. Fishbone double-layer barbed suture in cesarean section: a help in preventing long-term obstetric sequelae? Arch Gynecol Obstet. 2021 Sep;304(3):573-576. doi: 10.1007/s00404-021-06121-8. PMID 34146146
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581